CLINICAL TRIAL: NCT06142890
Title: Evaluating the Efficacy of Ceiling Fans for Limiting Heat Strain in Elderly Adults During Bed Rest in an Extreme Heat Event
Brief Title: Efficacy of Ceiling Fans for Mitigating Thermal Strain During Bed Rest in Older Adults During Heat Waves
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ottawa (Other)
Responsible Party: Principal Investigator, Glen P. Kenny, Full Professor, University of Ottawa
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: H-11-21-7575
Record Dates: First submitted 2023-11-13; First posted 2023-11-22 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Hyperthermia; Heat Stress; Cooling; Aging
Keywords: Heat wave; Cooling intervention; Elderly; Thermoregulation; Cardiovascular strain; Extreme heat event
MeSH Terms: conditions — Hyperthermia; Heat Stress Disorders

STUDY DESIGN:
Intervention Model Description: Each participant will complete 2 simulated heat wave exposures in random order: i) bed-rest; no fan cooling (control) and ii) bed-rest positioned beneath a ceiling fan providing standard air flow.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be informed of the study interventions before providing informed consent but will be masked to the order of the arms until exposure (i.e., participants will not know the fan conditions before entering the environmental chamber). Data will be blinded prior to analysis (including during statistical analysis).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No cooling intervention (control) (Active Comparator): Adults aged 65-85 years with or without type 2 diabetes and/or hypertension
  Interventions: Other: No cooling (control)
- Ceiling fan generating airflow (Experimental): Adults aged 65-85 years with or without type 2 diabetes and/or hypertension
  Interventions: Other: Cooling with ceiling fan

INTERVENTIONS:
Other: No cooling (control) — Participants are exposed to 31°C, 45% relative humidity for 8 hours without cooling intervention (control condition). Drinking water is available ad libitum. Participants remain in supine position with slight (~20°) chest and head elevation (low-Fowlers position) throughout the duration of bed-rest exposure.
  Arms: No cooling intervention (control)
Other: Cooling with ceiling fan — Participants are exposed to 31°C, 45% relative humidity for 8 hours. Drinking water is available ad libitum. Participants remain in supine position with slight (~20°) chest and head elevation (low-Fowlers position) throughout the duration of bed-rest exposure. Participants will remain under a commercially available ceiling fan generating a standard air flow throughout the duration of exposure.
  Arms: Ceiling fan generating airflow

SUMMARY:
With the increasing regularity and intensity of hot weather and heat waves, there is an urgent need to develop heat-alleviation strategies able to provide targeted protection for heat-vulnerable older adults. While air-conditioning provides the most effective protection from extreme heat, it is inaccessible for many individuals. Air-conditioning is also energy intensive, which can strain the electrical grid and, depending on the source of electricity generation, contribute to green house gas emissions. For these reasons, recent guidance has recommended the use of electric fans as a sustainable cooling alternative. While fans may increase sweat evaporation and heat loss in healthy, young adults, evidence supporting their use in older adults is scarce. Further, studies show that when environmental temperature exceeds skin temperature, fans are not effective and can even exacerbate hyperthermia in older adults. While older adults only account for ~13% of the population, they account for ~40% off all hospitalizations. In the context of sustainable cooling interventions, this is of particular importance given that many hospitals and long-term care homes do not have air-conditioning and rely on ceiling fans to enhance sweat evaporation while participants are bed-resting. While recent biophysical modelling has suggested that pedestal fans likely provide a clinically meaningful cooling effect (proposed to be ≥0.3°C) in temperatures below ~34°C in older adults, the efficacy of ceiling fans in mitigating heat strain in these conditions is currently unknown.

To address these knowledge gaps, this randomized crossover trial will evaluate body core temperature, cardiovascular strain, orthostatic intolerance, dehydration, and thermal comfort in adults aged 65-85 years exposed for 8-hours to conditions experienced during indoor overheating occurring during a heat wave in a temperate continental climate (31°C, 45% relative humidity). Each participant will complete two randomized exposures that will differ only in the airflow generated by a ceiling fan: no airflow (control) or standard airflow. Participants will remain in a supine position for the duration of the 8-hour exposure period, except for during hour 7 when they will complete a series of cardiovascular autonomic response tests.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults.
* Aged 65-85 years.
* Non-smoking.
* English or French speaking.
* Ability to provide informed consent.

Exclusion Criteria:

* Physical restriction (e.g., due to disease: intermittent claudication, renal impairment, active proliferative retinopathy, unstable cardiac or pulmonary disease, disabling stroke, severe arthritis, etc.).
* Use of or changes in medication judged by the patient or investigators to make participation in this study inadvisable (e.g., medications increasing risk of heat-related illness; beta blockers, anticholinergics, etc.)
* Cardiac abnormalities identified via 12-lead ECG during an incremental exercise test to volitional fatigue (performed for all participants).
* Peak aerobic capacity (VO2peak), as measured during an incremental exercise test to volitional fatigue, exceeding the 50th percentile of age- and sex-specific normative values published by the American College of Sports Medicine (ACSM).

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-12-05 (Actual); Primary Completion 2024-02-10 (Actual); Study Completion 2024-02-10 (Actual)

PRIMARY OUTCOMES:
Core temperature (peak) | End of heat exposure (hour 8)
  Peak rectal temperature (15 min average) during exposure. Rectal temperature is measured continuously throughout each simulated heat wave.

SECONDARY OUTCOMES:
Core temperature (AUC) | End of heat exposure (hour 8)
  Area under the curve of rectal temperature (in degree-hours).
Core temperature (end-exposure) | End of heat exposure (hour 8)
  Rectal temperature measured at hour 8 of the simulated heat wave exposure (15-min average)
Heart rate (peak) | End of heat exposure (hour 8)
  Peak heart rate (15 min average) during exposure. Heart rate is measured continuously via 3-lead ECG throughout each simulated heat wave
Heart rate (end-exposure) | End of heat exposure (hour 8)
  Heart rate measured at hour 8 of the simulated heat wave exposure (15-min average)
Heart rate (AUC) | End of heat exposure (hour 8)
  Area under the curve of rectal temperature (total beats).
Cardiac Response to Standing From Supine (30:15 Ratio) | During heat exposure (hour 7)
  Cardiac response to standing evaluated as the ratio between the highest R-wave to R-wave interval (lowest heart rate) measured at the 30th heart beat after standing from supine (+/- 5 beats) and the lowest R-wave to R-wave interval (highest heart rate) measured at the 15th heart beat after standing (+/- 5 beats). Cardiac response to standing will be evaluated twice, during two lying-to-standing tests (separated by 10 min of supine rest).
Systolic Response to Standing From Supine | During heat exposure (hour 7)
  Systolic blood pressure response to standing evaluated as the difference in blood pressure measured between the standing and supine. Standing systolic blood pressure will be taken as the lowest value of those measured after 60 and 120 seconds of standing. Systolic response to standing will be evaluated twice, during two lying-to-standing tests (separated by 10 min of supine rest).
Systolic blood pressure | End of heat exposure (hour 8)
  Systolic blood pressure measured in triplicate via automated oscillometry (~60 seconds between measures)
Diastolic blood pressure | End of heat exposure (hour 8)
  Diastolic blood pressure measured in triplicate via automated oscillometry (~60 seconds between measures)
Rate pressure product (end-exposure) | End of heat exposure (hour 8)
  Rate pressure product, an index of myocardial work and strain, calculated as systolic blood pressure x heart rate.
Heart rate variability: SDNN (end-exposure) | During heat exposure (hour 7)
  Standard deviation of normal-to-normal R-wave to R-wave intervals (SDNN) measured during 5 minutes of paced breathing (15 breaths/min) with participants in the seated position. SDNN will be evaluated twice, during two paced breathing periods (separated by 4 min of seated rest).
Heart rate variability: RMSSD (end-exposure) | During heat exposure (hour 7)
  Root mean squared standard deviation of normal-to-normal R-wave to R-wave intervals (RMSSD) measured during 5 minutes of paced breathing (15 breaths/min) with participants in the seated position. RMSSD will be evaluated twice, during two paced breathing periods (separated by 4 min of seated rest).
Fluid consumption | End of heat exposure (hour 8)
  Average hourly fluid consumption calculated by weighing participant water intake at the start and end of each hour of exposure (normalized to the exposure duration).
Whole-body sweat rate | End of heat exposure (hour 8)
  Average hourly whole-body sweat rate calculated as the change body mass during each exposure presented as a percentage of baseline body mass (corrected for food/water consumption and urination and normalized to the exposure duration)
Fluid loss | End of heat exposure (hour 8)
  Fluid loss calculated as the change in body mass during each exposure presented as a percentage of baseline body mass (corrected for food consumption)
Change in plasma volume | End of heat exposure (hour 8)
  Change in plasma volume from baseline values calculated from duplicate measurements of hemoglobin and hematocrit at the start and end of each exposure using the technique by Dill and Costill.
Thermal comfort scale (end-exposure) | End of heat exposure (hour 8)
  Thermal comfort assessed via a visual analog scale ("How comfortable does your body temperature feel?") ranging from "extremely uncomfortable" to "extremely comfortable"(midpoint: neutral).
Orthostatic intolerance symptoms assessment | During heat exposure (hour 7)
  Cumulative sum of scores on 6 questions asking participant to rank symptoms associated with orthostatic intolerance during the lying to standing tests. All symptoms scored on a scale from 0 (none) to 10 (worst possible) and include feelings of: (1) "dizziness, lightheadedness, feeling faint, or feeling like you might black out"; (2) "Problems with vision (blurring, seeing spots, tunnel vision, etc.)"; (3) "Weakness"; (4) "Fatigue"; (5) "Trouble concentrating"; and (6) "Head and neck discomfort".

CONTACTS AND LOCATIONS:
Overall Officials: Glen P Kenny, PhD, Principal Investigator — University of Ottawa
Locations (1):
- University of Ottawa, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participant data will be made available with approved analysis plan and signed access agreement
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Following publication of the main report(s)
Access Criteria: Approved analysis plan and signed access agreement

REFERENCES:
- [Derived] O'Connor FK, Meade RD, Janetos KT, Li-Maloney C, Sigal RJ, Boulay P, Kenny GP. Effect of Ceiling Fans on Core Temperature in Bed-Resting Older Adults Exposed to Indoor Overheating. J Am Geriatr Soc. 2026 Jan;74(1):200-204. doi: 10.1111/jgs.70109. Epub 2025 Sep 27. PMID 41014079